CLINICAL TRIAL: NCT01214421
Title: Multi-center, Open-label, Extension Study to Evaluate the Long-term Efficacy and Safety of Oral Tolvaptan Tablet Regimens in Subjects With Autosomal Dominant Polycystic Kidney Disease (ADPKD)
Brief Title: Tolvaptan Extension Study in Participants With ADPKD
Acronym: TEMPO 4/4
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 156-08-271; 2010-018401-10 (EudraCT Number)
Record Dates: First submitted 2010-09-26; First posted 2010-10-05 (Estimated); Results first posted 2021-10-25 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-09

CONDITIONS: Autosomal Dominant Polycystic Kidney Disease (ADPKD)
Keywords: Kidney Disease; ADPKD; Autosomal Dominant Polycystic Kidney Disease; Adult Polycystic Kidney Disease
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant; Kidney Diseases | interventions — Tolvaptan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tolvaptan (Experimental): Participants received a daily split-dose of tolvaptan titrated to the maximally tolerated dose, starting daily tolvaptan dose of 45 milligrams (mg) in the morning [AM]/15 mg in the evening [PM] titrated to 60 mg [AM]/30 mg [PM], then 90 mg [AM]/30 mg [PM] based on tolerability were given orally twice daily until the last participant originating from prior studies (either 156-04-251 or 156-04-250, 156-06-260, 156-09-284, 156-09-285, and 156-09-290) who was eligible for efficacy analysis completed the Month 24.
  Interventions: Drug: Tolvaptan

INTERVENTIONS:
Drug: Tolvaptan — Tablets of 15 or 30 mg
  Other Names: OPC-41061; Jinarc

SUMMARY:
To demonstrate whether tolvaptan modifies ADPKD progression as measured by changes from Baseline (from Study 156-04-251) in total kidney volume (TKV) and renal function.

ELIGIBILITY:
Inclusion Criteria:

- Participants who had successfully completed a Phase 1, 2, or 3 tolvaptan ADPKD or renal impairment study, with a confirmed diagnosis of ADPKD from prior studies [either 156-04-251 (NCT00428948) or 156-04-250 (NCT00413777), 156-06-260, 156-09-284 (NCT01336972), 156-09-285 (NCT01210560), and 156-09-290 (NCT01451827)].

Exclusion Criteria:

* Participants unable to provide written informed consent.
* Participants (men or women) would not adhere to the reproductive precautions as outlined in the Informed Consent Form.
* Participants (women only) with a positive urine pregnancy test.
* Participants who were pregnant or breast-feeding.
* Participants unable to take oral medications.
* Participants who had allergic reactions to tolvaptan or chemically related structures such as benzazepines (benzazepril, conivaptan, fenoldopam mesylate, or mirtazapine).
* Participants with disorders in thirst recognition or an inability to access fluids.
* Participants with critical electrolyte imbalances, as determined by the investigator
* Participants with or at risk of significant hypovolemia, as determined by investigator.
* Participants with significant anemia, as determined by investigator.
* Participants with a history of substance abuse (within the last 3 years).
* Participants who were taking other experimental (that is, non-marketed) therapies or were participating in another clinical drug or device study; participating in the off-drug follow-up period of another ADPKD trial with tolvaptan was permitted.
* Participants unable to complete magnetic resonance imaging (MRI) assessments (for example, participants with ferro-magnetic prostheses, aneurysm clips, severe claustrophobia).
* Participants who had taken a vasopressin antagonist (outside of previous participation in a tolvaptan study).
* Participants unable to comply with anti-hypertensive or other important medical therapy.
* Participants with advanced diabetes.
* Participants who were taking medications or had an illness that could confound endpoint assessments (including taking approved therapies for the purpose of affecting polycystic kidney disease [PKD] cysts).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1083 (Actual)
Dates: Start 2010-05-26 (Actual); Primary Completion 2016-02-29 (Actual); Study Completion 2016-02-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Otsuka Pharmaceutical Development & Commercialization, Inc.
Locations (89):
- United States (36):
  - Otsuka Investigational Site, Mobile, Alabama
  - Otsuka Investigational Site, Peoria, Arizona
  - Otsuka Investigational Site, Tempe, Arizona
  - Otsuka Investigational Site, Los Angeles, California
  - Otsuka Investigational Site, Palo Alto, California
  - Otsuka Investigational Site, San Diego, California
  - Otsuka Investigational Site, Aurora, Colorado
  - Otsuka Investigational Site, New Haven, Connecticut
  - Otsuka Investigational Site, Jacksonville, Florida
  - Otsuka Investigational Site, Port Charlotte, Florida
  - Otsuka Investigational Site, Atlanta, Georgia
  - Otsuka Investigational Site, Augusta, Georgia
  - Otsuka Investigational Site, Chicago, Illinois
  - Otsuka Investigational Site, Kansas City, Kansas
  - Otsuka Investigational Site, Baton Rouge, Louisiana
  - Otsuka Investigational Site, Baltimore, Maryland
  - Otsuka Investigational Site, Rockville, Maryland
  - Otsuka Investigational Site, Boston, Massachusetts
  - Otsuka Investigational Site, Detroit, Michigan
  - Otsuka Investigational Site, Minneapolis, Minnesota
  - Otsuka Investigational Site, Rochester, Minnesota
  - Otsuka Investigational Site, Voorhees Township, New Jersey
  - Otsuka Investigational Site, Buffalo, New York
  - Otsuka Investigational Site, Hawthorne, New York
  - Otsuka Investigational Site, New York, New York
  - Otsuka Investigational Site, Chapel Hill, North Carolina
  - Otsuka Investigational Site, Cincinnati, Ohio
  - Otsuka Investigational Site, Cleveland, Ohio
  - Otsuka Investigational Site, Portland, Oregon
  - Otsuka Investigational Site, Bethlehem, Pennsylvania
  - Otsuka Investigational Site, Philadelphia, Pennsylvania
  - Otsuka Investigational Site, Anderson, South Carolina
  - Otsuka Investigational Site, Nashville, Tennessee
  - Otsuka Investigational Site, Arlington, Texas
  - Otsuka Investigational Site, McAllen, Texas
  - Otsuka Investigational Site, Charlottesville, Virginia
- Argentina (4):
  - Otsuka Investigational Site, C.a.b.a., Buenos Aires
  - Otsuka Investigational Site, Pilar, Buenos Aires
  - Otsuka Investigational Site, Buenos Aires
  - Otsuka Investigational Site, Córdoba
- Australia (6):
  - Otsuka Investigational Site, St Leonards, New South Wales
  - Otsuka Investigational Site, Westmead, New South Wales
  - Otsuka Investigational Site, Woolloongabba, Queensland
  - Otsuka Investigational Site, Adelaide, South Australia
  - Otsuka Investigational Site, Parkville, Victoria
  - Otsuka Investigational Site, Perth, Western Australia
- Belgium (2):
  - Otsuka Investigational Site, Brussels
  - Otsuka Investigational Site, Ghent
- Canada (2):
  - Otsuka Investigational Site, Halifax, Nova Scotia
  - Otsuka Investigational Site, Montreal, Quebec
- France (7):
  - Otsuka Investigational Site, Bordeaux
  - Otsuka Investigational Site, Caen
  - Otsuka Investigational Site, Lyon
  - Otsuka Investigational Site, Paris
  - Otsuka Investigational Site, Reims
  - Otsuka Investigational Site, Saint-Etienne
  - Otsuka Investigational Site, Toulouse
- Germany (5):
  - Otsuka Investigational Site, Dresden
  - Otsuka Investigational Site, Düsseldorf
  - Otsuka Investigational Site, Essen
  - Otsuka Investigational Site, Heidelberg
  - Otsuka Investigational Site, Nuremberg
- Italy (5):
  - Otsuka Investigational Site, Bergamo
  - Otsuka Investigational Site, Milan
  - Otsuka Investigational Site, Modena
  - Otsuka Investigational Site, Napoli
  - Otsuka Investigational Site, Pavia
- Netherlands (2):
  - Otsuka Investigational Site, Amsterdam
  - Otsuka Investigational Site, Groningen
- Poland (7):
  - Otsuka Investigational Site, Ciechanów
  - Otsuka Investigational Site, Krakow
  - Otsuka Investigational Site, Lodz
  - Otsuka Investigational Site, Lublin
  - Otsuka Investigational Site, Szczecin
  - Otsuka Investigational Site, Warsaw
  - Otsuka Investigational Site, Wroclaw
- Romania (2):
  - Otsuka Investigational Site, Bucharest
  - Otsuka Investigational Site, Iași
- Russia (3):
  - Otsuka Investigational Site, Kemerovo
  - Otsuka Investigational Site, Saint Petersburg
  - Otsuka Investigational Site, Tomsk
- United Kingdom (8):
  - Otsuka Investigational Site, Belfast
  - Otsuka Investigational Site, Birmingham
  - Otsuka Investigational Site, Brighton
  - Otsuka Investigational Site, Coventry
  - Otsuka Investigational Site, Edinburgh
  - Otsuka Investigational Site, Inverness
  - Otsuka Investigational Site, London
  - Otsuka Investigational Site, Swansea

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available after marketing approval in global markets or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on the Vivli data sharing platform which can be found here: https://vivli.org/ourmember/Otsuka/
URL: https://clinical-trials.otsuka.com

REFERENCES:
- [Derived] Lioudis M, Zhou X, Davenport E, Nunna S, Krasa HB, Oberdhan D, Fernandes AW. Effects of tolvaptan discontinuation in patients with autosomal dominant polycystic kidney disease: a post hoc pooled analysis. BMC Nephrol. 2023 Jun 22;24(1):182. doi: 10.1186/s12882-023-03247-6. PMID 37349694
- [Derived] Chebib FT, Zhou X, Garbinsky D, Davenport E, Nunna S, Oberdhan D, Fernandes A. Tolvaptan and Kidney Function Decline in Older Individuals With Autosomal Dominant Polycystic Kidney Disease: A Pooled Analysis of Randomized Clinical Trials and Observational Studies. Kidney Med. 2023 Apr 14;5(6):100639. doi: 10.1016/j.xkme.2023.100639. eCollection 2023 Jun. PMID 37250503
- [Derived] Alpers DH, Lewis JH, Hunt CM, Freston JW, Torres VE, Li H, Wang W, Hoke ME, Roth SE, Westcott-Baker L, Estilo A. Clinical Pattern of Tolvaptan-Associated Liver Injury in Trial Participants With Autosomal Dominant Polycystic Kidney Disease (ADPKD): An Analysis of Pivotal Clinical Trials. Am J Kidney Dis. 2023 Mar;81(3):281-293.e1. doi: 10.1053/j.ajkd.2022.08.012. Epub 2022 Sep 30. PMID 36191725
- [Derived] Bennett H, McEwan P, Hamilton K, O'Reilly K. Modelling the long-term benefits of tolvaptan therapy on renal function decline in autosomal dominant polycystic kidney disease: an exploratory analysis using the ADPKD outcomes model. BMC Nephrol. 2019 Apr 23;20(1):136. doi: 10.1186/s12882-019-1290-5. PMID 31014270
- [Derived] Thimmappa ND, Blumenfeld JD, Cerilles MA, Dunning A, Donahue SL, Bobb WO, Zhang HL, Prince MR. Cisterna chyli in autosomal dominant polycystic kidney disease. J Magn Reson Imaging. 2015 Jan;41(1):142-8. doi: 10.1002/jmri.24527. Epub 2014 Jan 27. PMID 24470398
- [Derived] Blumenfeld JD, Tepler J, Mauer A, Coller B, Bichet DG, Smith B. Tolvaptan inhibition of desmopressin effects on coagulation factors in a patient with decreased von Willebrand factor and polycystic kidney disease. Blood. 2011 Jul 14;118(2):474-6. doi: 10.1182/blood-2011-04-347328. No abstract available. PMID 21757630

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 106 sites in 13 countries from 26 May 2010 to 29 Feb 2016. Eligible participants with autosomal dominant polycystic kidney disease (ADPKD) or renal impairment who completed previous tolvaptan treatment in studies: 156-04-251 (NCT00428948), 156-04-250 (NCT00413777), 156-06-260, 156-09-284 (NCT01336972), 156-09-285 (NCT01210560), and 156-09-290 (NCT01451827) were enrolled in this open-label study.
Pre-assignment Details: All enrolled participants received tolvaptan in this study. Data in this study was collected and reported as per the prior treatment received - tolvaptan (called as early treated) or placebo (called as delayed treated), for study 156-04-251 and all other studies combined.
Groups:
- Tolvaptan (From Study 156-04-251: Tolvaptan, Early Treated): Participants received a daily split-dose of tolvaptan titrated to the maximally tolerated dose, starting daily tolvaptan dose of 45 milligram (mg) in the morning [AM]/15 mg in the evening [PM] titrated to 60 mg [AM]/30 mg [PM], then 90 mg [AM]/30 mg [PM] based on tolerability were given orally twice daily up to Month 24. Participants were previously treated with tolvaptan in previous Study 156-04-251, hence called as Early Treated.
- Tolvaptan (From Study 156-04-251: Placebo, Delayed Treated): Participants received a daily split-dose of tolvaptan titrated to the maximally tolerated dose, starting daily tolvaptan dose of 45 mg [AM]/15 mg [PM] titrated to 60 mg [AM]/30 mg [PM], then 90 mg [AM]/30 mg [PM] based on tolerability were given orally twice daily up to Month 24. Participants were previously treated with placebo in the previous Study 156-04-251, hence called as Delayed Treated.
- Tolvaptan (From Other Studies: Tolvaptan, Early Treated): Participants received a daily split-dose of tolvaptan titrated to the maximally tolerated dose, starting daily tolvaptan dose of 45 mg [AM]/15 mg [PM] titrated to 60 mg [AM]/30 mg [PM], then 90 mg [AM]/30 mg [PM] based on tolerability were given orally twice daily up to Month 24. Participants were previously treated with tolvaptan in other studies (156-04-250, 156-06-260, 156-09-284, 156-09-285, and 156-09-290), hence called as Early Treated.
- Tolvaptan (From Other Studies: Placebo, Delayed Treated): Participants received a daily split-dose of tolvaptan titrated to the maximally tolerated dose, starting daily tolvaptan dose of 45 mg [AM]/15 mg [PM] titrated to 60 mg [AM]/30 mg [PM], then 90 mg [AM]/30 mg [PM] based on tolerability were given orally twice daily up to Month 24. Participants were previously treated with placebo in other studies (156-04-250, 156-06-260, 156-09-284, 156-09-285, and 156-09-290), hence called as Delayed Treated.
Period: Overall Study
Arm/Group | Tolvaptan (From Study 156-04-251: Tolvaptan, Early Treated) | Tolvaptan (From Study 156-04-251: Placebo, Delayed Treated) | Tolvaptan (From Other Studies: Tolvaptan, Early Treated) | Tolvaptan (From Other Studies: Placebo, Delayed Treated)
Started | 557 | 314 | 181 | 31
Completed | 507 | 256 | 143 | 22
Not Completed | 50 | 58 | 38 | 9
Not completed — Lost to Follow-up | 7 | 3 | 7 | 3
Not completed — Adverse Event | 16 | 35 | 14 | 3
Not completed — Sponsor Discontinued Site | 1 | 2 | 0 | 0
Not completed — Withdrawal Criteria Met | 3 | 0 | 2 | 1
Not completed — Physician Decision | 2 | 0 | 4 | 0
Not completed — Withdrawal by Subject | 21 | 18 | 11 | 2

BASELINE CHARACTERISTICS:
Population: The enrolled sample consisted of all participants who were enrolled in this open-label study.
Groups:
- Tolvaptan (From Study 156-04-251: Tolvaptan, Early Treated): Participants received a daily split-dose of tolvaptan titrated to the maximally tolerated dose, starting daily tolvaptan dose of 45 mg [AM]/15 mg [PM] titrated to 60 mg [AM]/30 mg [PM], then 90 mg [AM]/30 mg [PM] based on tolerability were given orally twice daily up to Month 24. Participants were previously treated with tolvaptan in previous Study 156-04-251, hence called as Early Treated.
- Total: Total of all reporting groups
Arm/Group | Tolvaptan (From Study 156-04-251: Tolvaptan, Early Treated) | Tolvaptan (From Study 156-04-251: Placebo, Delayed Treated) | Tolvaptan (From Other Studies: Tolvaptan, Early Treated) | Tolvaptan (From Other Studies: Placebo, Delayed Treated) | Total
Number analyzed (Participants) | 557 | 314 | 181 | 31 | 1083
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.2 (6.9) | 42.5 (7.2) | 40.0 (10.1) | 35.6 (8.7) | 41.7 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 254 | 156 | 91 | 15 | 516
  Male | 303 | 158 | 90 | 16 | 567
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 24 | 19 | 8 | 4 | 55
  Not Hispanic or Latino | 471 | 249 | 172 | 27 | 919
  Unknown or Not Reported | 62 | 46 | 1 | 0 | 109
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 535 | 302 | 169 | 27 | 1033
  Black/African American | 9 | 2 | 2 | 3 | 16
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1
  Asian | 3 | 2 | 5 | 0 | 10
  Other | 10 | 8 | 4 | 1 | 23

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From the Baseline in Total Kidney Volume (TKV) for Study 156-04-251 Participants Enrolled in This Study (156-08-271)
Description: Total kidney volume is a measure of disease progression in the ADPKD participants. Kidney volume was assessed in T1-weighted magnetic resonance images collected at each study site and sent to a central reviewing facility. At the central reviewing facility, radiologists used proprietary software to measure the volume of both kidneys in participants continuing from previous study (156-04-251) at Month 24 of this study (156-08-271) comparing change in TKV for the early-treated (those previously treated with tolvaptan) to delayed-treated (those previously treated with placebo). The percent change in the volume of both kidneys combined was analysed using mixed-effect model repeated measures (MMRM) analysis and reported. This outcome measure was analyzed only in the participants enrolled from the previous study - 156-04-251, as pre-specified in the protocol.
Time Frame: Study Baseline (Prior to Day 1 in Study 156-04-251) to Month 24 in this study (Study 156-08-271)
Population: The Efficacy Sample consisted of all enrolled participants who took at least 1 dose of study drug and completed 3 years of study drug treatment in previous Study 156-04-251. Overall number of participants analyzed signifies the number of participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- Tolvaptan, Early Treated (From Study 156-04-251: Tolvaptan): Participants received a daily split-dose of tolvaptan titrated to the maximally tolerated dose, starting daily tolvaptan dose of 45 mg [AM]/15 mg [PM] titrated to 60 mg [AM]/30 mg [PM], then 90 mg [AM]/30 mg [PM] based on tolerability were given orally twice daily up to Month 24. Participants were previously treated with tolvaptan in Study 156-04-251.
- Tolvaptan, Delayed Treated (From Study 156-04-251: Placebo): Participants received a daily split-dose of tolvaptan titrated to the maximally tolerated dose, starting daily tolvaptan dose of 45 mg [AM]/15 mg [PM] titrated to 60 mg [AM]/30 mg [PM], then 90 mg [AM]/30 mg [PM] based on tolerability were given orally twice daily up to Month 24. Participants were previously treated with placebo in Study 156-04-251.
Arm/Group | Tolvaptan, Early Treated (From Study 156-04-251: Tolvaptan) | Tolvaptan, Delayed Treated (From Study 156-04-251: Placebo)
Number analyzed (Participants) | 505 | 267
percent change | 28.66 (26.14) | 30.58 (27.21)
Statistical Analysis 1: Comparison: Tolvaptan, Early Treated (From Study 156-04-251: Tolvaptan) vs Tolvaptan, Delayed Treated (From Study 156-04-251: Placebo); Test type: Superiority; p = 0.358, Mixed Models Analysis; Ratio of geometric means (final values) = 0.99, 95% CI 2-sided [0.96 to 1.02]; Derived from the least squares (LS) mean difference between the treatment groups at each visit using MMRM model with factors of treatment, visit, region, baseline, baseline hypertensive status, baseline renal volume status, baseline creatinine clearance status, interaction of treatment and visit, and interaction of baseline and visit

2. Secondary Outcome: Change From the Baseline in Estimated Glomerular Filtration Rate (eGFR) as Assessed by Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) for Study 156-04-251 Participants Enrolled in This Study (156-08-271)
Description: Estimated Glomerular Filtration Rate (eGFR) according to CKD-EPI is calculated using the CKD-EPI equation, expressed as a single equation, is GFR = 141 × min (serum creatinine [Scr]/κ, 1)α × max(Scr/κ, 1)^-1.209 × 0.993 Age × 1.018 (if female) × 1.159 (if black), where Scr is serum creatinine, κ is 0.7 for females and 0.9 for males, α is -0.329 for females and -0.411 for males, min indicates the minimum of Scr/ĸ or 1, and max indicates the maximum of Scr/κ or 1 in participants continuing from previous study (156-04-251) at Month 24 of this study (156-08-271) comparing change in eGFR for the early-treated (those previously treated with tolvaptan) to delayed-treated (those previously treated with placebo). MMRM was used for the analysis. This outcome measure was analyzed only in the participants enrolled from the previous - 156-04-251, as pre-specified in the protocol.
Time Frame: Study Baseline (Prior to Day 1 in Study 156-04-251) to Month 24 in this study (Study 156-08-271)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Deviation); unit: mL/min/1.73 square meters (m^2)
Arm/Group | Tolvaptan, Early Treated (From Study 156-04-251: Tolvaptan) | Tolvaptan, Delayed Treated (From Study 156-04-251: Placebo)
Number analyzed (Participants) | 503 | 263
mL/min/1.73 square meters (m^2) | -16.77 (13.16) | -19.92 (16.40)
Statistical Analysis 1: Comparison: Tolvaptan, Early Treated (From Study 156-04-251: Tolvaptan) vs Tolvaptan, Delayed Treated (From Study 156-04-251: Placebo); Test type: Superiority; p = 0.0003, Mixed Models Analysis; LS mean difference (final values) = 3.15, 95% CI 2-sided [1.462 to 4.836]; Derived from MMRM analysis with fixed factors of treatment, visit, treatment visit interaction, hypertensive status, renal volume status and creatinine clearance status at baseline, region, baseline value, and baseline visit interaction as covariates, and with a heterogeneous toeplitz variance covariance matrix

3. Secondary Outcome: Annualized Slope of Total Kidney Volume (TKV) for Study 156-04-251 Participants Enrolled in Study 156-08-271
Description: Annualized slope of TKV is a measure of renal function and disease progression in ADPKD participants. The annualized slope is calculated as percentage of growth in TKV (measured in mL by MRI) divided by each participant's years of participation for all participants was calculated using MMRM analysis in participants continuing from previous study (156-04-251) at Month 24 of this study (156-08-271) comparing annualized slope of TKV for the early-treated (those previously treated with tolvaptan) to delayed-treated (those previously treated with placebo). This outcome measure was analyzed only in the participants enrolled from the previous study - 156-04-251, as pre-specified in the protocol.
Time Frame: Study Baseline (Prior to Day 1 in Study 156-08-271) to Month 24 in this study (Study 156-08-271)
Population: as for outcome 1
Measure: Number; unit: percent change in TKV/participant-years
Arm/Group | Tolvaptan, Early Treated (From Study 156-04-251: Tolvaptan) | Tolvaptan, Delayed Treated (From Study 156-04-251: Placebo)
Number analyzed (Participants) | 509 | 268
percent change in TKV/participant-years | 6.164 | 4.960
Statistical Analysis 1: Comparison: Tolvaptan, Early Treated (From Study 156-04-251: Tolvaptan) vs Tolvaptan, Delayed Treated (From Study 156-04-251: Placebo); Test type: Non-Inferiority — The non-inferiority for early-treatment and delayed-treatment groups; p = 0.0462, Mixed Models Analysis; Ratio of geometric means (final values) = 1.011, 95% CI 2-sided [1.000 to 1.023]; Derived from testing interaction of time and treatment using linear mixed model in which intercept and time are treated as random effects

4. Secondary Outcome: Annualized Slope of eGFR (CKD-EPI) for Study 156-04-251 Participants Enrolled in Study 156-08-271
Description: Annualized slope of eGFR (CKD-EPI) is a measure of renal function and disease progression in ADPKD participants. The annualized slope of eGFR (CKD-EPI) (divided by each participant's years of participation) for all participants was calculated using MMRM analysis in participants continuing from previous study (156-04-251) at Month 24 of this study (156-08-271) comparing change in TKV for the early-treated (those previously treated with tolvaptan) to delayed-treated (those previously treated with placebo). eGFR was calculated using the Chronic Kidney Disease-Epidemiology (CKD-EPI) formula. This outcome measure was analyzed only in the participants enrolled from the previous study - 156-04-251, as pre-specified in the protocol.
Time Frame: Study Baseline (Prior to Day 1 in Study 156-08-271) to Month 24 (Study 156-08-271)
Population: as for outcome 1
Measure: Number; unit: ml/min/1.73m^2/participant-years
Arm/Group | Tolvaptan, Early Treated (From Study 156-04-251: Tolvaptan) | Tolvaptan, Delayed Treated (From Study 156-04-251: Placebo)
Number analyzed (Participants) | 549 | 304
ml/min/1.73m^2/participant-years | -3.255 | -3.142
Statistical Analysis 1: Comparison: Tolvaptan, Early Treated (From Study 156-04-251: Tolvaptan) vs Tolvaptan, Delayed Treated (From Study 156-04-251: Placebo); Test type: Non-Inferiority — The non-inferiority for early-treatment and delayed-treatment groups; p = 0.7259, Mixed Models Analysis; Ratio of geometric means (final values) = -0.113, 95% CI 2-sided [-0.746 to 0.520]; [other analysis details as in outcome 3, analysis 1]

5. Secondary Outcome: Annualized TKV Slope for Study 156-04-251 Placebo Participants Enrolled in Study 156-08-271
Description: Annualized slope of TKV is a measure of renal function and disease progression in ADPKD participants. The annualized slope is calculated as percentage of growth in TKV (measured in mL by MRI) divided by each participant's years of participation, using MMRM analysis to compare annualized slope of TKV for the participants who received placebo in previous study (156-04-251) to annualized slope of TKV for the same participants who received tolvaptan in this study (156-08-271). This outcome measure was analyzed only in the participants enrolled from the previous study - 156-04-251 and who received placebo in the previous study, as pre-specified in the protocol.
Time Frame: Tolvaptan, Delayed Treated: Baseline to Month 24 in Study 156-08-271; Placebo: Baseline to Month 36 in Study 156-04-251
Population: as for outcome 1
Measure: Number; unit: percent change in TKV/participant-years
Groups:
- Tolvaptan, Delayed Treated (In Study 156-08-271): Participants received a daily split-dose of tolvaptan titrated to the maximally tolerated dose, starting daily tolvaptan dose of 45 mg [AM]/15 mg [PM] titrated to 60 mg [AM]/30 mg [PM], then 90 mg [AM]/30 mg [PM] based on tolerability were given orally twice daily up to Month 24. Participants were previously treated with placebo in Study 156-04-251.
- Placebo (In Study 156-04-251): Participants were treated with placebo in the previous Study 156-04-251.
Arm/Group | Tolvaptan, Delayed Treated (In Study 156-08-271) | Placebo (In Study 156-04-251)
Number analyzed (Participants) | 268 | 268
percent change in TKV/participant-years | 4.779 | 5.627
Statistical Analysis 1: Comparison: Tolvaptan, Delayed Treated (In Study 156-08-271) vs Placebo (In Study 156-04-251); Test type: Superiority; p = 0.1080, Mixed Models Analysis; Ratio of geometric means (final values) = 0.992, 95% CI 2-sided [0.982 to 1.002]; Derived from linear mixed model with terms of participant, treatment, time, interaction of treatment and time, interaction of participant and time, and baseline for intra-participant comparison between 251 and 271. Time and intercept are treated as random effects

6. Secondary Outcome: Annualized Slope of Renal Function (eGFRCKD-EPI) for Study 156-04-251 Placebo Participants Enrolled in Study 156-08-271
Description: Annualized slope of eGFR (CKD-EPI) is a measure of renal function and disease progression in ADPKD participants. The annualized slope of eGFR (calculated using CKD-EPI formula) divided by each participant's years of participation, using MMRM analysis to compare annualized slope of eGFR (CKD-EPI) for the participants who received placebo in previous study (156-04-251) to the annualized slope of eGFR (CKD-EPI) for the same participants who received tolvaptan in this study (156-08-271). This outcome measure was analyzed only in the participants enrolled from the previous study - 156-04-251 who received placebo in previous study and received tolvaptan in this study, as pre-specified in the protocol.
Time Frame: Tolvaptan, Delayed Treated: Baseline to Month 24 in Study 156-08-271; Placebo: Baseline to Month 36 in Study 156-04-251
Population: as for outcome 1
Measure: Number; unit: ml/min/1.73m^2/participant-years
Arm/Group | Tolvaptan, Delayed Treated (In Study 156-08-271) | Placebo (In Study 156-04-251)
Number analyzed (Participants) | 304 | 304
ml/min/1.73m^2/participant-years | -3.211 | -3.572
Statistical Analysis 1: Comparison: Tolvaptan, Delayed Treated (In Study 156-08-271) vs Placebo (In Study 156-04-251); Test type: Superiority; p = 0.2265, Mixed Models Analysis; Ratio of geometric means (final values) = 0.361, 95% CI 2-sided [-0.224 to 0.946]; [other analysis details as in outcome 5, analysis 1]

ADVERSE EVENTS:
Time Frame: From the signing of the informed consent form until the end of the study regardless of whether the participants were on or off active study medication (Up to approximately 5 years)
Arm/Group | Tolvaptan (From Study 156-04-251: Tolvaptan, Early Treated) | Tolvaptan (From Study 156-04-251: Placebo, Delayed Treated) | Tolvaptan (From Other Studies: Tolvaptan, Early Treated) | Tolvaptan (From Other Studies: Placebo, Delayed Treated)
All-Cause Mortality (participants affected / at risk) | 5/557 | 0/314 | 0/181 | 0/31
Serious Adverse Events (participants affected / at risk) | 143/557 | 79/314 | 34/181 | 5/31
Other Adverse Events (participants affected / at risk) | 528/557 | 310/314 | 175/181 | 29/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tolvaptan (From Study 156-04-251: Tolvaptan, Early Treated) (N=557) | Tolvaptan (From Study 156-04-251: Placebo, Delayed Treated) (N=314) | Tolvaptan (From Other Studies: Tolvaptan, Early Treated) (N=181) | Tolvaptan (From Other Studies: Placebo, Delayed Treated) (N=31)
Anaemia (Blood and lymphatic system disorders) | 2 | 1 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Accelerated Idioventricular Rhythm (Cardiac disorders) | 0 | 0 | 0 | 1
Acute Coronary Syndrome (Cardiac disorders) | 1 | 1 | 0 | 0
Acute Myocardial Infarction (Cardiac disorders) | 1 | 1 | 0 | 0
Angina Pectoris (Cardiac disorders) | 0 | 0 | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 2 | 2 | 0 | 0
Bradycardia (Cardiac disorders) | 2 | 0 | 0 | 0
Cardiac Arrest (Cardiac disorders) | 1 | 0 | 1 | 0
Coronary Artery Disease (Cardiac disorders) | 1 | 1 | 0 | 0
Myocardial Infarction (Cardiac disorders) | 3 | 0 | 0 | 0
Myocardial Ischaemia (Cardiac disorders) | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0
Pericarditis (Cardiac disorders) | 2 | 1 | 0 | 0
Prinzmetal Angina (Cardiac disorders) | 0 | 1 | 0 | 0
Sinus Arrhythmia (Cardiac disorders) | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Congenital Cystic Kidney Disease (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Goitre (Endocrine disorders) | 1 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0 | 0
Cataract (Eye disorders) | 1 | 1 | 0 | 0
Retinal Detachment (Eye disorders) | 0 | 1 | 0 | 0
Abdominal Hernia (Gastrointestinal disorders) | 1 | 2 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 2 | 0 | 0
Abdominal Pain Lower (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Gastritis Erosive (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Ileus Paralytic (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Inguinal Hernia (Gastrointestinal disorders) | 5 | 3 | 0 | 0
Intestinal Fistula (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Large Intestine Polyp (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Localised Intraabdominal Fluid Collection (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Pancreatitis Acute (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Pancreatitis Necrotising (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Umbilical Hernia (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Peripheral Swelling (General disorders) | 0 | 0 | 1 | 0
Systemic Inflammatory Response Syndrome (General disorders) | 0 | 0 | 1 | 0
Bile Duct Stone (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Biliary Dyskinesia (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 2 | 0 | 0
Cholecystitis Acute (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Drug-Induced Liver Injury (Hepatobiliary disorders) | 0 | 2 | 0 | 0
Haemorrhagic Hepatic Cyst (Hepatobiliary disorders) | 1 | 0 | 0 | 1
Hepatic Cyst (Hepatobiliary disorders) | 4 | 0 | 0 | 0
Hepatic Failure (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hepatic Pain (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hepatocellular Injury (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Portal Hypertension (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Allergy to Arthropod Sting (Immune system disorders) | 0 | 1 | 0 | 0
Atopy (Immune system disorders) | 1 | 0 | 0 | 0
Drug Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0
Abdominal Abscess (Infections and infestations) | 1 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0
Bronchopulmonary Aspergillosis (Infections and infestations) | 0 | 1 | 0 | 0
Catheter Site Infection (Infections and infestations) | 0 | 1 | 0 | 0
Cervicitis (Infections and infestations) | 0 | 0 | 1 | 0
Chronic Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0
Clostridium Difficile Colitis (Infections and infestations) | 1 | 0 | 0 | 0
Clostridium Difficile Infection (Infections and infestations) | 1 | 0 | 0 | 0
Diarrhoea Infectious (Infections and infestations) | 1 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 2 | 1 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis Viral (Infections and infestations) | 0 | 0 | 2 | 0
Genital Herpes (Infections and infestations) | 1 | 0 | 0 | 0
Kidney Infection (Infections and infestations) | 1 | 1 | 0 | 0
Lobar Pneumonia (Infections and infestations) | 2 | 0 | 0 | 0
Mastitis (Infections and infestations) | 1 | 0 | 0 | 0
Pharyngitis Streptococcal (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Pulmonary Tuberculosis (Infections and infestations) | 1 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 6 | 1 | 2 | 0
Renal Cyst Infection (Infections and infestations) | 9 | 3 | 2 | 0
Sepsis (Infections and infestations) | 3 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 1 | 0 | 1
Ureteritis (Infections and infestations) | 0 | 0 | 1 | 0
Urinary Tract Infection (Infections and infestations) | 4 | 1 | 0 | 0
Urosepsis (Infections and infestations) | 1 | 1 | 1 | 0
Viral Pericarditis (Infections and infestations) | 1 | 0 | 0 | 0
Wound Infection (Infections and infestations) | 1 | 0 | 0 | 0
Accidental Overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Expired Product Administered (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Femur Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Gun Shot Wound (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Incisional Hernia (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Joint Dislocation (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Ligament Rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Ligament Sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Limb Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Meniscus Injury (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Renal Haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Shunt Occlusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Tendon Rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Alanine Aminotransferase Increased (Investigations) | 2 | 3 | 5 | 1
Aspartate Aminotransferase Increased (Investigations) | 1 | 1 | 3 | 1
Blood Alkaline Phosphatase Increased (Investigations) | 0 | 1 | 0 | 0
Blood Bilirubin Increased (Investigations) | 0 | 0 | 1 | 0
Blood Creatine Phosphokinase Increased (Investigations) | 0 | 0 | 1 | 0
Blood Creatinine Increased (Investigations) | 6 | 6 | 1 | 0
Blood Lactate Dehydrogenase Increased (Investigations) | 0 | 0 | 0 | 1
Gamma-Glutamyltransferase Increased (Investigations) | 0 | 3 | 0 | 0
Glomerular Filtration Rate Decreased (Investigations) | 1 | 0 | 0 | 0
Haemoglobin Decreased (Investigations) | 1 | 0 | 0 | 0
Hepatic Enzyme Increased (Investigations) | 0 | 1 | 0 | 0
Liver Function Test Abnormal (Investigations) | 1 | 2 | 0 | 0
Smear Cervix Abnormal (Investigations) | 1 | 0 | 0 | 0
Transaminases Increased (Investigations) | 3 | 2 | 2 | 0
Vasopressin Challenge Test Abnormal (Investigations) | 0 | 0 | 1 | 0
White Blood Cell Count Increased (Investigations) | 0 | 0 | 1 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Chondropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Flank Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Foot Deformity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0
Loose Body In Joint (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0
Cervix Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Cholesterin Granuloma Of Middle Ear (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Endometrial Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Gastrointestinal Stromal Tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Intraductal Proliferative Breast Lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0
Plasma Cell Myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Testis Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 1 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 1 | 0 | 0
Carotid Artery Aneurysm (Nervous system disorders) | 1 | 0 | 0 | 0
Carotid Artery Dissection (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebral Atrophy (Nervous system disorders) | 0 | 1 | 0 | 0
Cerebrovascular Accident (Nervous system disorders) | 1 | 3 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0
Essential Tremor (Nervous system disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 1 | 0
Intracranial Aneurysm (Nervous system disorders) | 3 | 3 | 1 | 0
Ischaemic Stroke (Nervous system disorders) | 0 | 1 | 0 | 0
Lumbar Radiculopathy (Nervous system disorders) | 0 | 1 | 0 | 0
Occipital Neuralgia (Nervous system disorders) | 1 | 0 | 0 | 0
Polyneuropathy (Nervous system disorders) | 1 | 0 | 0 | 0
Subarachnoid Haemorrhage (Nervous system disorders) | 2 | 0 | 0 | 0
Transient Ischaemic Attack (Nervous system disorders) | 2 | 0 | 0 | 0
Ectopic Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0
Gestational Hypertension (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 1 | 0 | 0
Major Depression (Psychiatric disorders) | 1 | 0 | 0 | 0
Suicide Attempt (Psychiatric disorders) | 1 | 0 | 0 | 0
Acute Kidney Injury (Renal and urinary disorders) | 2 | 3 | 1 | 0
Calculus Ureteric (Renal and urinary disorders) | 0 | 0 | 1 | 0
Calculus Urinary (Renal and urinary disorders) | 1 | 0 | 0 | 0
Chronic Kidney Disease (Renal and urinary disorders) | 5 | 2 | 2 | 0
Haematuria (Renal and urinary disorders) | 1 | 1 | 0 | 0
Nephropathy (Renal and urinary disorders) | 0 | 1 | 0 | 0
Renal Cyst (Renal and urinary disorders) | 2 | 1 | 0 | 0
Renal Cyst Haemorrhage (Renal and urinary disorders) | 6 | 4 | 2 | 0
Renal Cyst Ruptured (Renal and urinary disorders) | 1 | 1 | 0 | 0
Renal Failure (Renal and urinary disorders) | 2 | 0 | 1 | 0
Renal Haemorrhage (Renal and urinary disorders) | 1 | 0 | 0 | 0
Renal Impairment (Renal and urinary disorders) | 6 | 3 | 1 | 0
Renal Pain (Renal and urinary disorders) | 1 | 2 | 0 | 0
Urinary Incontinence (Renal and urinary disorders) | 0 | 1 | 0 | 0
Urine Flow Decreased (Renal and urinary disorders) | 1 | 0 | 0 | 0
Breast Discomfort (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Breast Haematoma (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Endometriosis (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Postmenopausal Haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Acute Lung Injury (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Nasal Septum Deviation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pharyngeal Oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Hidradenitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Aneurysm (Vascular disorders) | 1 | 0 | 0 | 0
Aortic Dissection (Vascular disorders) | 1 | 0 | 0 | 0
Arterial Stenosis (Vascular disorders) | 1 | 0 | 0 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 1 | 0 | 0
Peripheral Arterial Occlusive Disease (Vascular disorders) | 0 | 1 | 0 | 0
Peripheral Venous Disease (Vascular disorders) | 0 | 1 | 0 | 0
Subclavian Vein Thrombosis (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tolvaptan (From Study 156-04-251: Tolvaptan, Early Treated) (N=557) | Tolvaptan (From Study 156-04-251: Placebo, Delayed Treated) (N=314) | Tolvaptan (From Other Studies: Tolvaptan, Early Treated) (N=181) | Tolvaptan (From Other Studies: Placebo, Delayed Treated) (N=31)
Anaemia (Blood and lymphatic system disorders) | 35 | 20 | 13 | 0
Abdominal Pain (Gastrointestinal disorders) | 37 | 15 | 13 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 23 | 16 | 4 | 0
Constipation (Gastrointestinal disorders) | 23 | 25 | 8 | 1
Diarrhoea (Gastrointestinal disorders) | 60 | 30 | 13 | 2
Dry Mouth (Gastrointestinal disorders) | 45 | 44 | 25 | 4
Dyspepsia (Gastrointestinal disorders) | 29 | 15 | 8 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 24 | 11 | 10 | 2
Nausea (Gastrointestinal disorders) | 42 | 32 | 22 | 2
Vomiting (Gastrointestinal disorders) | 32 | 15 | 9 | 2
Fatigue (General disorders) | 53 | 54 | 32 | 2
Oedema Peripheral (General disorders) | 51 | 32 | 9 | 1
Thirst (General disorders) | 261 | 161 | 80 | 13
Bronchitis (Infections and infestations) | 30 | 17 | 4 | 1
Gastroenteritis (Infections and infestations) | 31 | 20 | 9 | 2
Gastroenteritis Viral (Infections and infestations) | 12 | 7 | 6 | 2
Influenza (Infections and infestations) | 42 | 25 | 18 | 1
Nasopharyngitis (Infections and infestations) | 83 | 55 | 18 | 4
Sinusitis (Infections and infestations) | 40 | 19 | 13 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 61 | 35 | 28 | 2
Urinary Tract Infection (Infections and infestations) | 61 | 33 | 16 | 4
Aspartate Aminotransferase Increased (Investigations) | 19 | 5 | 7 | 2
Blood Creatinine Increased (Investigations) | 96 | 39 | 20 | 2
Decreased Appetitie (Metabolism and nutrition disorders) | 5 | 13 | 12 | 1
Gout (Metabolism and nutrition disorders) | 35 | 9 | 6 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 37 | 15 | 2 | 2
Polydipsia (Metabolism and nutrition disorders) | 62 | 51 | 38 | 6
Vitamin D Deficiency (Metabolism and nutrition disorders) | 34 | 16 | 13 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 57 | 16 | 13 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 60 | 40 | 15 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 28 | 18 | 5 | 1
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 38 | 11 | 7 | 2
Dizziness (Nervous system disorders) | 30 | 36 | 13 | 1
Headache (Nervous system disorders) | 75 | 56 | 20 | 2
Haematuria (Renal and urinary disorders) | 47 | 36 | 13 | 4
Nocturia (Renal and urinary disorders) | 145 | 111 | 94 | 17
Pollakiuria (Renal and urinary disorders) | 30 | 24 | 20 | 4
Polyuria (Renal and urinary disorders) | 231 | 175 | 111 | 22
Renal Cyst Ruptured (Renal and urinary disorders) | 3 | 2 | 2 | 3
Renal Pain (Renal and urinary disorders) | 147 | 90 | 43 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 42 | 23 | 10 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 7 | 12 | 7 | 3
Hypertension (Vascular disorders) | 160 | 82 | 42 | 2

LIMITATIONS AND CAVEATS:
The trial did not meet its primary endpoint as both groups showed similar decreases in the rate of TKV growth due in part to unforeseen limitations in the trial design. However, early-treatment resulted in cumulative improvements in renal function.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right to review results publications prior to public release and can delay such publications for a period greater than 60 days but no more than 120 days from the date that the publication is submitted to the Sponsor for review. Sponsor can require changes to the publication to protect Sponsor's intellectual property rights and/or confidential information and reserves the right to limit publication timing and scope of data published based on the number of study locations.